CLINICAL TRIAL: NCT03014011
Title: Effects of Mild Hypoglycaemia on Cognitive Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); Psychiatric Centre Rigshospitalet (Other)
Responsible Party: Principal Investigator, Malin Nilsson, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MISP
Record Dates: First submitted 2016-12-21; First posted 2017-01-09 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type II; Hypoglycemia; Cognitive Change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Glucose Clamp Technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoglycaemic clamp first, then euglyceamic clamp (Other): First intervention with a hypoglycaemic clamp (one examination day of approximately 5 hours), there after a wash out period of 21-42 days, then second and final intervention day with an euglycaemic clamp (approximately 5 hours).
  Interventions: Other: Hypoglycaemic clamp; Other: Euglycaemic clamp
- Euglycaemic clamp first, then hypoglycaemic clamp (Other): First intervention with an euglycaemic clamp (one examination day of approximately 5 hours), there after a wash out period of 21-42 days, then second and final intervention day with a hypoglycaemic clamp (approximately 5 hours).
  Interventions: Other: Hypoglycaemic clamp; Other: Euglycaemic clamp

INTERVENTIONS:
Other: Hypoglycaemic clamp — The clamp is performed by insulin and adjustable 20% glucose infusions, with the aim to lower and keep plasma blood glucose levels at 3 mmol/L for outcome measurements.
Other: Euglycaemic clamp — The clamp is performed by insulin and adjustable 20% glucose infusions, with the aim to keep plasma blood glucose levels at 6 mmol/L for outcome measurements.

SUMMARY:
Hypoglycaemia in subjects suffering from type 2 diabetes may have substantial consequences including a significant negative impact on quality of life. Further, repeated minor hypoglycaemias may result in significant productivity losses.

Here, the investigators propose to provide quantitative results on cognition during an acute mild hypoglycaemic episode (target plasma glucose 3 mmol/L) in 28 subjects with type 2 diabetes. Data will be provided on executive function, attention and memory.

DETAILED DESCRIPTION:
Hypoglycaemia in subjects suffering from type 2 diabetes may have substantial consequences including a significant negative impact on quality of life. Further, repeated minor hypoglycaemias may result in significant productivity losses. In healthy subjects a number of studies show that during a hypoglycaemic episode with plasma levels of 2.2 - 2.5 mmol/L (40-45 mg/dl) brain areas responsible for cognition have an altered neuronal function when measuring cerebral blood flow. This is accompanied by severely impaired cognitive function with a reduced ability to solve simple cognitive tasks. At higher levels of glucose (above 3 mmol/L (54 mg/dl)), it remains to be settled whether cognitive functions are also affected negatively and whether this may be accompanied by changes in brain metabolism. Apart from raising the blood glucose directly or indirectly via glucagon, no treatment for hypoglycaemia exists, but since Glucagon-like peptide-1 (GLP-1) based therapies used in type 2 diabetes may affect brain glucose consumption, therapeutic interventions to prevent negative results of hypoglycaemia may eventually become clinically possible.

Here, the investigators propose to provide quantitative results on cognition during an acute mild hypoglycaemic episode (target plasma glucose 3 mmol/L). Data will be provided on executive function, attention and memory.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent
* Clinically diagnosed type 2 diabetes mellitus for at least 3 months (diagnosed according to the criteria of the World Health Organization (WHO)).
* Normal haemoglobin ≥ 8.0 mmol/L (male) or ≥ 6.4 mmol/L (female)
* Male or female participants aged 35-70 years, both inclusive.
* Treated with diet or any antidiabetic medication except sulfonylureas, meglitinides or insulin.
* HbA1c ≤ 9.0 % by local laboratory analysis.
* BMI >23 kg/m2 and <35 kg/m2

Exclusion Criteria:

* Receipt of any investigational medicinal product within 3 months before screening in this trial.
* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder.
* Nephropathy (serum creatinine levels ≥ 126 μmol/L (male) or ≥ 111 μmol/L (female)).
* Cardiac problems defined as decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time and/or angina pectoris within the last 12 months and/or acute myocardial infarction at any time.
* Active or recent malignant disease.
* Treatment with drugs that cannot be paused for 12 hours.
* Repeated resting blood pressure at screening outside the range 90-140 mmHg for systolic or 50-90 mmHg for diastolic. This exclusion criterion also pertains to subjects taking antihypertensives.
* Visual impairment or auditory impairment.
* Known abnormalities of the central nervous system or any endocrinological (with the exception of diabetes mellitus and euthyroid goiter), haematological, neurological, psychiatric diseases or other major disorders that in the opinion of the investigator precludes compliance with the protocol, evaluation of the results or represent an unacceptable risk for the participant's safety.
* Proliferative retinopathy (funduscopy performed within 3 months before the screening is acceptable) and/or severe neuropathy.
* Current treatment with systemic drugs, which may interfere with glucose metabolism.
* Significant history of alcoholism or drug/chemical abuse as per investigator's judgement.
* Current tobacco user (smoking or nicotinic product use 3 months prior to screening).
* Severe hypoglycaemic event during the past 6 months.
* Known hypoglycaemia unawareness.
* Participants with mental incapacity or language barriers precluding adequate understanding or co-operation or who, in the opinion of the investigator or their general practitioner, should not participate in the trial.
* For females only: Pregnancy, breast-feeding status or intention of becoming pregnant during the trial.
* Any chronic disorder or severe disease that in the opinion of the investigator might endanger participant's safety or compliance with the protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Rungby, Professor, Principal Investigator — Department of Endocrinology, Bispebjerg University Hospital, Denmark
Locations (1):
- Department of Research in Endocrinology, Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson M, Jensen N, Gejl M, Bergmann ML, Storgaard H, Zander M, Miskowiak K, Rungby J. Experimental non-severe hypoglycaemia substantially impairs cognitive function in type 2 diabetes: a randomised crossover trial. Diabetologia. 2019 Oct;62(10):1948-1958. doi: 10.1007/s00125-019-4964-4. Epub 2019 Jul 31. PMID 31367958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 participants were screened between May 2017 and July 2018 at the Department of Endocrinology, Bispebjerg University Hospital, Denmark.
Pre-assignment Details: Of the 37 screened participants, 28 met inclusion criteria and were randomised. 25 completed both intervention visits. Three participants (one man, two women) withdrew from the study after randomisation for reasons not related to the intervention. Baseline characteristics are based on the 25 participants that completed the study.
Groups:
- Hypoglycaemic Clamp Followed by Euglycaemic Clamp: Participants completed a hypoglycaemic clamp on a first intervention visit. After a washout period of at least 2 weeks (maximum of 6 weeks), a euglycaemic clamp was performed on the second intervention visit.
- Euglycaemic Clamp Followed by Hypoglycaemic Clamp: Participants completed a euglycaemic clamp on a first intervention visit. After a washout periodof at least 2 weeks (maximum of 6 weeks), a hypoglycaemic clamp was performed on the second intervention visit.
Period: First Intervention
Arm/Group | Hypoglycaemic Clamp Followed by Euglycaemic Clamp | Euglycaemic Clamp Followed by Hypoglycaemic Clamp
Started (Participants randomized and started intervention visit) | 14 | 13
Completed (Participants who completed the intervention visit) | 13 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout
Arm/Group | Hypoglycaemic Clamp Followed by Euglycaemic Clamp | Euglycaemic Clamp Followed by Hypoglycaemic Clamp
Started (started intervention visit) | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Hypoglycaemic Clamp Followed by Euglycaemic Clamp | Euglycaemic Clamp Followed by Hypoglycaemic Clamp
Started | 12 | 13
Completed (completed intervention visit) | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Randomised, double-blinded, crossover study design
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 25

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Speed
Description: Symbol Digit Modalities Test was used as a measurement of psychomotor speed.
  For the Symbol Digit Modalities Test, participants were required to use a coded key to match nine abstract symbols paired with numerical digits. The final score is the correct number of substitutions in 120 s, and scores range between 0 and 110. Higher values represent a better outcome.
Time Frame: All neurocognitive testing was assessed at each intervention when glucose levels had been stabile for 40 minutes, an average of 2 hours after clamp procedure start. The duration of neurocognitive testing was approximately 40 min.
Population: The two interventions were hypoglycaemia (aiming for a plasma glucose target of 3.0 ± 0.2 mmol/l) and euglycaemia (plasma glucose clamp target 6.0 ± 0.2 mmol/l).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Hypoglycaemia: low glucose level
- Euglycaemia: normal glucose level
Arm/Group | Hypoglycaemia | Euglycaemia
Number analyzed (Participants) | 25 | 25
score on a scale | 48.7 (9.8) | 56.6 (12)

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was collected from the day they were included, until the day after their second (and final) intervention visit, an average of 2 months.
Groups:
- Hypoglycaemic Clamp: Mean plasma glucose concentration during the neurocognitive testing was 3.13 mmol/l for the hypoglycaemic clamp.
- Euglycaemic Clamp: Mean plasma glucose concentration during the neurocognitive testing was 5.83 mmol/l for the euglycaemic clamp.
Arm/Group | Hypoglycaemic Clamp | Euglycaemic Clamp
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03014011/Prot_SAP_000.pdf